CLINICAL TRIAL: NCT07403591
Title: Efficacy and Neural Mechanisms of Neuroimage-guided Dual-target Continuous Theta Burst Stimulation (Auditory Cortex and M1) for Generalized Anxiety Disorder
Brief Title: Mapsd Dual-target cTBS (Auditory Cortex and M1) for Generalized Anxiety Disorder
Acronym: Dual-ACM1-GAD
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Anhui Medical University (Other)
Responsible Party: Principal Investigator, WANG KAI, Professor, Anhui Medical University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: AHMU-GAD-Dual-ACM1-2026
Record Dates: First submitted 2026-02-04; First posted 2026-02-11 (Actual); Last update posted 2026-02-11 (Actual); Status verified 2026-02

CONDITIONS: Generalized Anxiety Disorder
Keywords: Generalized Anxiety Disorder; Continuous Theta Burst Stimulation; Transcranial Magnetic Stimulation; Neuronavigation; Dual-target; Auditory Cortex; Primary Motor Cortex
MeSH Terms: conditions — Generalized Anxiety Disorder

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Active Dual-target cTBS (Experimental): Participants will receive active continuous Theta Burst Stimulation (cTBS) guided by a neuronavigation system. The stimulation targets are the left auditory association cortex followed by the primary motor cortex (M1). Treatment will be administered three times a day for seven consecutive days.
  Interventions: Device: Active Dual-target cTBS
- Sham Dual-target cTBS (Sham Comparator): Participants will undergo a sham cTBS procedure using a placebo coil. The procedure mimics the sound, sensation, and coil placement (dual-target) of the active group but delivers no effective magnetic field.
  Interventions: Device: Sham Dual-target cTBS

INTERVENTIONS:
Device: Active Dual-target cTBS — A non-invasive brain stimulation technique using a MagStim Rapid2 stimulator with a 70mm air-cooled figure-of-eight coil.
  Targets: 1. Left auditory association cortex (MNI: -62, -40, 10), located using Brainsight neuronavigation. 2. Primary Motor Cortex (M1), determined by the resting motor threshold (RMT) hotspot. Protocol: Stimulation of the auditory cortex is immediately followed by M1 stimulation. Each target receives a standard cTBS protocol (3-pulse 50 Hz bursts repeated at 5 Hz, total 600 pulses, 40s duration). Dosing: Delivered at 100% RMT. Sessions are repeated 3 times/day with 15-min intervals for 7 days.
  Arms: Active Dual-target cTBS
Device: Sham Dual-target cTBS — A placebo procedure using an inert sham coil that is identical in appearance and sound to the active coil but does not deliver a significant magnetic field to the cortex. Blinding: The procedure includes identical neuronavigation setup, dual-target coil positioning (Auditory Cortex then M1), duration, and treatment schedule (3 times/day for 7 days) to maintain the blind.
  Arms: Sham Dual-target cTBS

SUMMARY:
The purpose of this study is to investigate the effectiveness of a dual-target non-invasive brain stimulation technique called continuous Theta Burst Stimulation (cTBS) for treating Generalized Anxiety Disorder (GAD). The researchers will use a neuronavigation system, which acts like a GPS for the brain, to guide the stimulation to two specific targets: the left auditory association cortex and the primary motor cortex (M1).

Participants will be randomly assigned to one of two groups. One group will receive active dual-target cTBS treatment, while the other will receive a sham (placebo) stimulation that feels similar but has no therapeutic effect. The treatment will be given three times a day for seven consecutive days. Before and after the treatment period, all participants will complete clinical questionnaires to measure their anxiety and undergo Magnetic Resonance Imaging (MRI) scans to help researchers understand how cTBS affects brain activity.

DETAILED DESCRIPTION:
This study is a randomized, triple-blind, sham-controlled trial designed to evaluate the efficacy and neural mechanisms of neuronavigation-guided dual-target continuous Theta Burst Stimulation (cTBS) in patients with Generalized Anxiety Disorder (GAD).

A total of participants diagnosed with GAD according to the Diagnostic and Statistical Manual of Mental Disorders, 5th Edition (DSM-5) will be recruited. After providing informed consent, participants will be randomized in a 1:1 ratio to receive either active dual-target cTBS or sham cTBS.

The active intervention involves stimulating two sequential targets using a MagStim Rapid2 stimulator with a 70mm air-cooled figure-of-eight coil:

Target 1 (Auditory Cortex): The first target is the left auditory association cortex (posterior superior temporal sulcus), located using a Brainsight neuronavigation system based on individual MRI scans transformed from MNI coordinates (-62, -40, 10).

Target 2 (M1): The second target is the primary motor cortex (M1), located at the site where the resting motor threshold (RMT) is determined.

Stimulation of the auditory cortex target will be immediately followed by stimulation of the M1 target. The cTBS protocol for each target consists of 3-pulse bursts at 50 Hz, repeated at a 5 Hz frequency, for a total of 600 pulses (40 seconds duration) per target. The stimulation intensity will be set at 100% of the individual's RMT. To achieve cumulative aftereffects, this dual-target protocol will be repeated three times per day with 15-minute intervals between sessions, for seven consecutive days.

The sham intervention will utilize an identical-looking sham coil that produces similar sounds and scalp sensations without inducing a significant magnetic field. The procedure, including neuronavigation, coil placement, and duration, is identical to the active group to maintain the triple-blind design (masking for participants, investigators, and outcomes assessors).

All participants will undergo comprehensive assessments at baseline, post-intervention, and follow-up. Assessments include clinical scales such as the Hamilton Anxiety Rating Scale (HAMA) and multimodal MRI (structural, rs-fMRI, and DTI) to examine neural network dynamics.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosis of Generalized Anxiety Disorder (GAD) according to the Diagnostic and Statistical Manual of Mental Disorders, 5th Edition (DSM-5), confirmed by at least two psychiatrists.
2. Hamilton Anxiety Rating Scale (HAMA) score > 14.
3. Age between 18 and 60 years.
4. Right-handed.
5. More than 5 years of education.
6. Patients are either medication-free or maintain a consistent medication regimen during cTBS treatment.
7. Willing and able to provide written informed consent.
8. Normal or corrected-to-normal visual acuity and hearing.

Exclusion Criteria:

1. Presence of other psychiatric disorders, such as substance abuse, schizophrenia, schizoaffective disorder, hysteria, autism, or bipolar disorder.
2. History of epilepsy, seizures, or severe neurological diseases (e.g., stroke, organic brain lesions).
3. Presence of severe somatic diseases, such as severe heart, liver, or renal insufficiency.
4. Pregnant or lactating women.
5. Contraindications to Transcranial Magnetic Stimulation (TMS) or Magnetic Resonance Imaging (MRI), such as the presence of a cardiac pacemaker, cochlear implant, cerebrovascular metal stent, or metal dentures.
6. Inability to cooperate with experimental procedures due to conditions such as severe claustrophobia.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2026-03-01 (Estimated); Primary Completion 2027-03-01 (Estimated); Study Completion 2027-04-01 (Estimated)

PRIMARY OUTCOMES:
Change from Baseline in Hamilton Anxiety Rating Scale (HAMA) Score | Baseline (Day 1), Post-intervention (Day 9), and 2-week Follow-up
  The HAMA is a 14-item, clinician-administered scale used to assess the severity of anxiety symptoms. Total scores range from 0 to 56, with higher scores indicating more severe anxiety. The change in total score from baseline to post-intervention and follow-up will be assessed.
Change from Baseline in Resting-State Neural Activity | Baseline (Day 1) and Post-intervention (Day 9)
  Changes in resting-state brain activity will be measured by functional magnetic resonance imaging (fMRI). Analyses will examine neural activity (ALFF/ReHo) and functional connectivity dynamics related to the stimulation targets (left auditory cortex and M1) and brain circuits implicated in anxiety.

SECONDARY OUTCOMES:
Change from Baseline in Hamilton Depression Rating Scale (HAMD-17) Score | Baseline (Day 1) and Post-intervention (Day 9)
  The HAMD-17 is a 17-item, clinician-rated scale to assess the severity of depression. Total scores range from 0 to 52, with higher scores indicating more severe depression.
Change from Baseline in Self-Rating Anxiety Scale (SAS) Score | Baseline (Day 1), Post-intervention (Day 9), and 2-week Follow-up
  The SAS is a 20-item self-report scale designed to measure the severity of anxiety symptoms. The standard score ranges from 25 to 100, where higher scores indicate more severe levels of anxiety.
Change from Baseline in Patient Health Questionnaire-15 (PHQ-15) Score | Baseline (Day 1) and Post-intervention (Day 9)
  The PHQ-15 is a 15-item self-report scale to assess the severity of somatic symptoms. Total scores range from 0 to 30, with higher scores indicating more severe somatic symptoms.
Change from Baseline in Pittsburgh Sleep Quality Index (PSQI) Score | Baseline (Day 1) and Post-intervention (Day 9)
  The PSQI is a self-report questionnaire assessing sleep quality. The global score ranges from 0 to 21, with higher scores indicating worse sleep quality.

CONTACTS AND LOCATIONS:
Locations (1):
- Anhui Medical University, Hefei, Anhui, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Neri F, Cappello C, Viberti F, Donniacuo A, Burzi L, Cinti A, Benelli A, Luca Smeralda C, Romanella S, Santarnecchi E, Mandala M, Rossi S. rTMS of the auditory association cortex improves speech intelligibility in patients with sensorineural hearing loss. Clin Neurophysiol. 2024 Apr;160:38-46. doi: 10.1016/j.clinph.2024.02.007. Epub 2024 Feb 9. PMID 38395005